CLINICAL TRIAL: NCT00729534
Title: Research Participant Perception of Care Project: Part 1: Focus Groups of Research Participants and Research Professionals to Identify Key Dimensions of the Research Participant Experience
Brief Title: Research Participants Perceptions of Their Experience in Clinical Studies
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080193; 08-CC-0193
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-05-29

CONDITIONS: Participant Satisfaction
Keywords: Perception; Focus Group; Perception of Clinical Research Participation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine how research volunteers experience their participation in studies in order to develop surveys to be used by research centers trying to improve the experience of their participants.

People 18 years of age and older who have participated in an NIH research protocol within the past 2 years as someone with a medical condition under study may be eligible for this study.

Eight participants will participate in a moderator facilitated focus group in a discussion about being in research studies. An observer audiotapes the discussion and takes written notes. The focus group discussion lasts about 1 to 1 (Omega) hours.

DETAILED DESCRIPTION:
The conduct of high quality clinical research is dependent on the ability to recruit and retain subjects who are invested in, understand, and have confidence in the clinical research process. Understanding subjects experiences as research volunteers is critical to the continual improvement of the processes of clinical research and, subsequently, to enhancing the subject s experience. Heretofore, studies evaluating the subject s comprehension of the informed consent process have served as, at best, an indirect measure of the quality of the subject s experience. Few, if any, studies have assessed the quality and efficacy of the entire clinical research process from the subject s perspective. This study is the first phase of a two-part study designed to directly measure research participants perceptions of all aspects of the clinical research process (e.g., recruitment, informed consent, education, autonomy and subject's rights, provision of clinical care) for the purposes of improving the clinical research subject s experience.

Obtaining robust, validated data requires a partnership between those with expertise in the design and analysis of surveys, and those who can articulate the needs of research participants and improve the way in which clinical research is conducted. For the former, we will be greatly advantaged by our partnership with NRC Picker, which has committed the resources necessary to assist the survey project development; conduct the focus groups, telephone interviews, and expert advisory group sessions required to further optimize the survey; collaborate in the analysis; and fund the second-stage formal validation of the survey. For the latter, we have assembled a collaborative team of research professionals from the CTSA award recipient centers, and interested GCRCs, with expertise in human subject protections, research ethics, research conduct, education and performance improvement.

The current study entails the recruitment and conduct of up to a total of 22 Focus Groups, each consisting of either 8-10 research subjects (12-16 groups) or 6-10 research professionals (6 groups), in order achieve the first goal: to assess the key dimensions of the research experience upon which to test the second part of the research, a perception of the research experience survey. The current study will involve 8-11 academic medical centers, enrolling a total of 100-128 research subjects, and 45-60 research professionals in total. A second goal of the project is to describe the process, obstacles and successes of implementing a multi-center protocol across the GCRCs and the CTSA consortium. A subsequent research protocol will concern the fielding and validation of that survey in approximately 3,700 subjects at up to 10 academic medical centers (CTSA and GCRC awardees).

ELIGIBILITY:
* INCLUSION CRITERIA:

You may be eligible to participate in this study if you:

* Are at least 18 years old.
* Are able to give informed consent.
* Have participated in an NIH research study within the past 2 years as someone with a medical condition under study.
* Can participate constructively and non-disruptively in the group discussion, in the opinion of the investigator.
* Are fluent in English

EXCLUSION CRITERIA:

You will not be able to be in this study if you:

* Do not sign the informed consent form.
* Do not agree to honor the confidentiality of others in the focus group.
* Do not agree to be recorded on audiotape.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08-01; Study Completion 2013-05-29

PRIMARY OUTCOMES:
To identify key dimensions of the clinical research process that influence participants' perception of their experience as a study participant

SECONDARY OUTCOMES:
To describe the process, obstacles and successes of implementing a multi-center protocol across the GCRCs and the CTSA consortium.

CONTACTS AND LOCATIONS:
Overall Officials: David K Henderson, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States